CLINICAL TRIAL: NCT06392984
Title: Ultrasonographic Measurement of Diaphragmatic Thickness in Adolescents With Pectus Deformity: Is it an Early Predictor of Respiratory Dysfunction?
Brief Title: Ultrasonographic Measurement of Diaphragmatic Thickness in Adolescents With Pectus Deformity
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 98
Record Dates: First submitted 2024-03-30; First posted 2024-05-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pectus Deformity; Pectus Excavatum; Pectus Carinatum; Pectus Abnormalities
Keywords: Pectus Deformity; Pectus Abnormalities; Diaphragma Thickness; Ultrasonographic Measurement
MeSH Terms: conditions — Funnel Chest; Pectus Carinatum | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants aged 6-18 years who were diagnosed with pectus deformity: Pectus deformity study form consisting of clinical and radiological measurements of participants aged 6-18 years who were diagnosed with pectus deformity and applied to the scoliosis outpatient clinic will be filled in detail.
  Interventions: Diagnostic Test: Pectus deformity study form; Diagnostic Test: Pulmonary function test; Diagnostic Test: Ultrasonographic Diaphragm Thickness Measurement
- Control group: Pectus deformity study form consisting of clinical and radiological measurements of participants aged 6-18 years who were diagnosed with normal and applied to the scoliosis outpatient clinic will be filled in detail.
  Interventions: Diagnostic Test: Pectus deformity study form; Diagnostic Test: Pulmonary function test; Diagnostic Test: Ultrasonographic Diaphragm Thickness Measurement

INTERVENTIONS:
Diagnostic Test: Pectus deformity study form — Pectus deformity study form consisting of clinical and radiological measurements of participants aged 6-18 years who applied to the outpatient clinic with chest deformity will be filled in detail.
Diagnostic Test: Pulmonary function test — Pulmonary function tests (PFTs) are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange. This information can help your healthcare provider diagnose and decide the treatment of certain lung disorders. Investigators will use handheld spirometry device for measurement. Three measurements will be made. In these three measurements; FEV1(Forced Expiratory Volume In One Second) (Liter-L), FEV1 (%predicted), FVC (Forced Vital Capacity) (Liter-L), FVC (%predicted), FEV1/FVC (%) and FEV1/FVC (%predicted) will be evaluated. The arithmetic average of the results of these three measurements will be taken.
  Other Names: • Spirometry Function Test
Diagnostic Test: Ultrasonographic Diaphragm Thickness Measurement — Diaphragm thickness (millimeter-mm) will be measured in the supine position with a 6-14 Mhz lineer, conventional ultrasound probe (Mindray DC-8, Shenzen Mindray Bio-Medical Electronics CO. LTD.,P.R. China) at the end of inspiration and expiration from the intercostal space on the anterior axillary line. The measurements will be evaluated by making three measurements from the right 8-9. intercostal space where the diaphragm is best visualized. End-expiratory (Forced residual capacity-FRC) (millimeter-mm), end-inspiratory (Total Lung Capacity-TLC) (millimeter-mm)) and thickening rate (%) (thickness TLC / thickness FRC) will be evaluated three times and the arithmetic average of these three measurements will be taken.

SUMMARY:
Pectus deformities are among the most common anterior chest wall pathologies. Pectus excavatum is the most common chest deformity with an incidence of 0.1-0.3%. In severe deformities, a decrease in lung volume is observed. This can cause decreased pulmonary function and affect the function of the right ventricle. The diaphragm is the main respiratory muscle, and diaphragm contraction is associated with respiratory functions. So, investigators aimed to measure diaphragmatic thickness in adolescents with pectus deformity and to show whether diaphragmatic thickness is an early predictor of respiratory disorder in participants who do not show any clinical symptoms or whose respiratory functions are normal.

DETAILED DESCRIPTION:
Pectus deformities are among the most common anterior chest wall pathologies. Pectus excavatum is the most common chest deformity with an incidence of 0.1-0.3%. It is more common in boys than girls at a ratio of 4:1. This deformity involves the lower part of the body of the sternum; The chest wall has shifted posteriorly.

Pectus excavatum is a cosmetic defect that in most cases does not have physiological consequences. In severe deformities, a decrease in lung volume is observed. This can cause decreased pulmonary function and affect the function of the right ventricle. Funnel chest defects can cause chest pain, shortness of breath, decreased cardiac output, and decreased exercise capacity, depending on the depth of the deformity.

The alignment of the skeletal system in the chest and its harmony with the compliance of the chest wall are related to respiratory function; changes in the rib cage lead to a decrease in lung capacity. The diaphragm is the main respiratory muscle, and diaphragm contraction is associated with respiratory functions. In recent years, ultrasonography (USG) has gained increasing utility for visualizing the diaphragm and assessing its function, with several advantages.

Based on this, investigators aimed to measure diaphragmatic thickness in adolescents with pectus deformity and to show whether diaphragmatic thickness is an early predictor of respiratory disorder in participants who do not show any clinical symptoms or whose respiratory functions are normal.

ELIGIBILITY:
Inclusion Criteria:

* Increased thoracal kyphosis (thoracic hyperkyphosis)
* Being between the ages of 6-18
* Patients who can cooperate with spirometry.

Exclusion Criteria:

* Congenital spinal, costal and diaphragmatic anomalies
* Neuromuscular disease
* Respiratory system diseases that affect lung functions
* Patients who cannot cooperate with spirometry.
* Having surgery to the chest wall or spine

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: It will consist of participants with pectus deformity who apply to the Physical Medicine and Rehabilitation Clinic of the University of Health Sciences Gaziosmanpaşa Training and Research Hospital within the study date ranges, meet the inclusion and exclusion criteria and voluntarily agree to participate in the research. Healthy individuals identical in age and gender will be included in the study as a control group. Demographic information of all individuals involved in the recruitment will be collected.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Pectus deformity study form | Within 1 month of applying to the outpatient clinic
  Pectus deformity study form consisting of clinical and radiological measurements of patients aged 6-18 years who applied to the outpatient clinic with chest deformity will be filled in detail.
Pulmonary function test | Within 1 month of applying to the outpatient clinic
  We will use handheld spirometry device for measurement. Three measurements will be made. In these three measurements; FEV1(Forced Expiratory Volume In One Second)(Liter-L), FEV1 (%predicted), FVC (Forced Vital Capacity) (Liter-L), FVC (%predicted), FEV1/FVC (%) and FEV1/FVC (%predicted) will be evaluated. The arithmetic average of the results of these three measurements will be taken.
Ultrasonographic Diaphragm Thickness Measurement | Within 1 month of applying to the outpatient clinic
  Diaphragm thickness (millimeter-mm) will be measured in the supine position with a 6-14 Mhz lineer, conventional ultrasound probe (Mindray DC-8, Shenzen Mindray Bio-Medical Electronics CO. LTD.,P.R. China) at the end of inspiration and expiration from the intercostal space on the anterior axillary line. The measurements will be evaluated by making three measurements from the right 8-9. intercostal space where the diaphragm is best visualized. End-expiratory (Forced residual capacity-FRC) (millimeter-mm), end-inspiratory (Total Lung Capacity-TLC) (millimeter-mm) and thickening rate (%) (thickness TLC / thickness FRC) will be evaluated three times and the arithmetic average of these three measurements will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Guneser Gulec, MD, Study Chair — Gaziosmanpasa Training and Research Hospital Physical Rehabilitation Department; Cansu Ozkan, MD, Study Chair — Medical Park Bahcelievler Hospital Physical Medicine and Rehabilitation Department
Locations (1):
- Zeynel Karakullukcuoglu,, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

REFERENCES:
- [Result] Ramadan S, Wilde J, Tabard-Fougere A, Toso S, Beghetti M, Vallee JP, Corbelli R, Barazzone-Argiroffo C, Lascombes P, Ruchonnet-Metrailler I. Cardiopulmonary function in adolescent patients with pectus excavatum or carinatum. BMJ Open Respir Res. 2021 Jul;8(1):e001020. doi: 10.1136/bmjresp-2021-001020. PMID 34326157
- [Result] Tomaszewski R, Wiktor L, Machala L. Evaluation of thoracic vertebrae rotation in patients with pectus excavatum. Acta Orthop Traumatol Turc. 2017 Jul;51(4):284-289. doi: 10.1016/j.aott.2017.03.005. Epub 2017 Jun 16. PMID 28624480
- [Result] Azimi G, Bozorgmehr R, Sattari P, Azimi A, Azimi H, Marzban-Rad S. Physiologic function of mediastinum space. Ann Med Surg (Lond). 2022 Sep 15;82:104670. doi: 10.1016/j.amsu.2022.104670. eCollection 2022 Oct. PMID 36268434